CLINICAL TRIAL: NCT04210973
Title: Efficacy and Safety Study of Anyu Peibo in the Treatment of Major Depressive Disorder(MDD): a Ⅲ Randomized, Double-Blind, Placebo-Paralleled, Multicenter Clinical Trial
Brief Title: Comparison of Anyu Peibo With Placebo in Treatment of MDD in China
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Su Zhou YiHua Biotechnology Co. LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AYPB-MDD-Ⅲ-201901; 2018ZX09734-005 (Other Grant/Funding Number: China National Major Project for IND)
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anyu Peibo (Experimental): Anyu Peibo Capsule, oral, 0.8g twice per day
  Interventions: Drug: Anyu Peibo
- Placebo (Placebo Comparator): Placebo,oral, twice per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anyu Peibo — Anyu Peibo Capsule, 0.8g twice per day, oral after breakfast and supper
  Arms: Anyu Peibo
Drug: Placebo — Placebo Capsule, twice per day, oral after breakfast and supper
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Anyu Peibo Capsule comparing with placebo in the treatment of Chinese Patients with Depression.

ELIGIBILITY:
Inclusion Criteria:

* Adult with primary diagnosis of major depressive disorder(MDD) based on the criteria of DSM-5, single episode or recurrent episode. [296.21; 296.22; 296.23; 296.31; 296.32; 296.33]
* The total score of MADRS is ≥26 in both screening visit and baseline visit.
* The first item of MADRS is ≥3 in both screening visit and baseline visit.
* CGI-S is ≥4 in both screening visit and baseline visit.
* The subject understands and consents to takes part in this clinical trials. The subjects should sign informed consent form.

Exclusion Criteria:

* The subject has a current psychiatric diagnosis other than depression.
* The subject has a suicide attempt within recent 1 year, or has a currently significant risk of suicide, or has a score ≥3 on item 10 (suicidal ideation) of MADRS.
* The subject has a current depressive episode due to somatic general disease or a neurological disease, such as hypothyroidism.
* When the MADRS total score of baseline visit compares with the screening visit, the decreasing rate is ≥25%.
* Known hypersensitivity to Big Leaf Ju, or at least to two kinds of drugs.
* Any unstable cardiovascular, hepatic, renal, blood, endocrine, or other medical disease.
* Any neurological disease (such as Parkinson's Disease, cerebrovascular accident and epilepsy) or cerebral injury (traumatic or disease related).
* Had a history or a high risk related disease or medication of seizure disorder, except infantile febrile convulsion.
* The subject could not take medication or has a disease affecting drug absorption, distribution, metabolism and excretion.
* Clinically significant electrocardiographic(ECG) abnormalities in screening visit. Such as QTc ≥450 ms in male or ≥470 ms in female.
* Clinically significant abnormal laboratory values (eg. ALT or AST value above 2 times of clinical top-limit; Cr value above normal top-limit; thyroid gland function index (≥ 2 items in 5 items) above 1.2 times or below 0.8 times of the normal range, or investigator diagnosed with hypothyroidism or hyperthyroidism).
* The subject who used at least two different antidepressants with recommended dose and adequate duration (maximum dosage by at least 4 weeks according to label) treatment still had no respond.
* The subject uses antidepressant drug normally before 2 weeks of screening, and stops using psychotropic drug before randomization less than 5 half-life period (monoamine oxidase inhibitor: at least 2 weeks; fluoxetine: at least 1 month).
* The subject received systematic light therapy, laser therapy and acupuncture or other Traditional Chinese Medicine, or systemic biofeedback therap within 2 weeks.
* The subject received modified ECT, trans-cranial magnetic stimulation (TMS), vagus nerve stimulation (VNS) or systematic psychotherapy within 3 months.
* Women who were pregnant, breast-feeding, or serum-HCG(+) on screening; or planning to become pregnant within 3 months after kick-off of clinical trial.
* Education level below junior high school.
* The subject has participated in a drug clinical trial within 1 month before screening.
* The investigator thinks the subject is unsuitable to enroll in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The change of total score from baseline in Montgomery Asberg Depression Rating Scale （MADRS） | 8 weeks
  the minimum and maximum values of MADRS are from 0 to 60, and higher scores mean a worse outcome

SECONDARY OUTCOMES:
Clinical Remission Rate according to total score of MADRS at the end of study | 8 weeks
  Remission=at the end of study, total score of MADRS ≤10, the minimum and maximum values of MADRS are from 0 to 60, and higher scores mean a worse outcome
Clinical Remission Rate according to 17-items Hamilton Depression Scale (HAMD17) total score at the end of study | 8 weeks
  Remission=at the end of study, total score of HAMD17 ≤7, the minimum and maximum values of HAMD17 are from 0 to 52, and higher scores mean a worse outcome
The change of total score of MADRS by time | 8 weeks
  the minimum and maximum values of MADRS are from 0 to 60, and higher scores mean a worse outcome
The change of total score from baseline in HAMD17 | 8 weeks
  the minimum and maximum values of HAMD17 are from 0 to 52, and higher scores mean a worse outcome
The change of total score from baseline in Hamilton Anxiety Scale (HAMA) | 8 weeks
  the minimum and maximum values of HAMA are from 0 to 56, and higher scores mean a worse outcome
The change of score from baseline in Clinical Global Impression-Severity of Illness (CGI-S) | 8 weeks
  the minimum and maximum values of CGI-S are from 1 to 7, and higher scores mean a worse outcome
Clinical Global Impression-Severity of Illness (CGI-I) score | 8 weeks
  the minimum and maximum values of CGI-I are from 1 to 7, and higher scores mean a worse outcome
The change of total score from baseline in Discriminative Scale Space Tracker (DSST) | 8 weeks
  the minimum and maximum values of DSST are from 0 to 90, and higher scores mean a better outcome
The change of total score from baseline in Trail Making Test (TMT) A&B | 8 weeks
  the minimum and maximum values of TMT are from 0 to 300, and higher scores mean a worse outcome
The change of total score from baseline in Sheehan Disability Scale (SDS) | 8 weeks
  the minimum and maximum values of SDS are from 0 to 10, and higher scores mean a worse outcome
Proportion of subjects who withdrew from clinical trial due to poor efficacy | 8 weeks
  Investigator will assess subject's efficacy according to his/her clinical status with rating scales, including MADRS, HAMD17, HAMA and CGI, which already listed in Outcome
Proportion of subjects who combined medication to treat insomnia | 8 weeks
Incidence rate of AE | 8 weeks
  AE=Adverse Events
Breath Rate | 8 weeks
  per minutes
Pulse Rate | 8 weeks
  per minutes
Heartbeat Rate | 8 weeks
  per minutes
Diastolic blood pressure | 8 weeks
  Sitting position, mmHg
Systolic blood pressure | 8 weeks
  Sitting position, mmHg
Electrocardiogram(ECG) | 8 weeks
  the number of subjects with abnormal ECG report by 12-lead electrocardiogram
Assessment of Arizona Sexual Experience Scale (ASES) | 8 weeks
  the minimum and maximum values of ASES are from 1 to 6, and higher scores mean a worse outcome
Number of Participants with AE result in early withdrawal from clinical trials | 8 weeks
Number of Participants with Serious Adverse Event (SAE) result in early withdrawal from clinical trials | 8 weeks
Number of Emerging AE during drug withdrawal period | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Huafang LI, MD. PhD., Principal Investigator — Shanghai Mental Health Center
Locations (15):
- China (15):
  - Beijing Anding Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Chongqing Mental Health Center, Chongqing, Chongqing Municipality
  - Guangzhou Brain Hospital, Guangzhou, Guangdong
  - The Sixth People's Hospital of Hebei Province, Baoding, Hebei
  - The Second Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Zhumadian mental Hospital, Zhumadian, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Jiangxi Mental Hospital, Nanchang, Jiangxi
  - Brain Hospital of Jilin Province, Siping, Jilin
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - XI'AN Mental Health Center, Xi’an, Shanxi
  - Ningbo Kangning Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang J, Yu Y, Jiang Y, Chen W, Li Y, Shen Y, Zheng Q, Li H. The efficacy and safety of Anyu Peibo Capsule in the treatment of patients with major depressive disorder in China: study protocol for a randomized placebo-controlled trial. Trials. 2021 Sep 3;22(1):585. doi: 10.1186/s13063-021-05550-9. PMID 34479619
- See also: EMEA :Guideline on clinical investigation of medicinal products in the treatment of depression. — https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-clinical-investigation-medicinal-products-treatment-depression_en.pdf
- See also: FDA.Major Depressive Disorder：Developing Drug for Treatment Guidance for Industry. — https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM611259.pdf